CLINICAL TRIAL: NCT05302739
Title: The Effects of Facial Cooling on Physiological and Perceptual Responses During Simulated Competition in Male Epee Fencers
Brief Title: The Effects of Facial Cooling on Fencing Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: StMarysUC3
Record Dates: First submitted 2022-03-04; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Hyperthermia
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facial cooling (Experimental): Between each simulated fencing match participants will spend the first 30 s of rest having a facial water mist sprayed onto the face with accompanying fanning from 50 cm away from the face.
  Interventions: Other: Facial cooling
- Placebo (No Intervention)

INTERVENTIONS:
Other: Facial cooling — 30 s of water mist sprayed onto the face during breaks in a simulated fencing competition
  Arms: Facial cooling

SUMMARY:
Fencing competitions can last between nine and eleven hours, during which athletes wear layers of protective equipment that impair evaporative heat transfer and spend a large amount of time at exercise intensities > 85% maximum heart rate. Fencing performance can potentially contribute to heat stress due to increases in core temperature. Elevated core temperatures could hamper performance, and therefore the implementation of a strategy to reduce core temperature increases could lead to augmented fencing performance. Cooling methods are limited for use between fencing matches and during short breaks within a direct elimination match. Furthermore, due to multiple layers of thick protective equipment cooling method applications are limited primarily to the facial area. A potential cooling strategy, during fencing competition, includes the utilization of a water facial mist spray combined with fanning of the face. Therefore, the aim of this study is to investigate the novel use of facial cooling on core temperature, relevant physiological parameters, perceived exertion and thermal comfort and sensation during a simulated fencing competition performance, in male epee fencers.

ELIGIBILITY:
Inclusion Criteria:

* Trained fencers

Exclusion Criteria:

* Injured or a contraindicative medical condition

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04-20 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-26 (Estimated)

PRIMARY OUTCOMES:
Tympanic temperature | From baseline to completion, up to 31 days
  Change from baseline in tympanic temperature taken during each 60 s break within the simulated fencing bout protocol and between each simulated fencing bout
Heart rate | From baseline to completion, up to 31 days
  Change from baseline in heart rate recorded during each 60 s break within the simulated fencing bout protocol and between each simulated fencing bout
Blood lactate concentration | From baseline to completion, up to 31 days
  Change from baseline in blood lactate concentration recorded during each 60 s break within the simulated fencing bout protocol and between each simulated fencing bout
Thermal comfort | From baseline to completion, up to 31 days
  Change from baseline in thermal comfort will be recorded on a scale of 1 - 4 (1 = comfortable; 2 = slightly uncomfortable; 3 = uncomfortable; 4 = very uncomfortable) during each 60 s break within the simulated fencing bout protocol and between each simulated fencing bout.
Thermal sensation | From baseline to completion, up to 31 days
  Change from baseline in thermal sensation will be recorded on a scale of 1 - 7 (1 = cold; 2 = cool; 3 = slightly cool; 4 = neutral; 5 = slightly warm; 6 = warm; 7 = hot) during each 60 s break within the simulated fencing bout protocol and between each simulated fencing bout.
Rating of perceived exertion of the dominant arm | From baseline to completion, up to 31 days
  Change from baseline in rating of perceived exertion exertion for the dominant arm will be recorded on a scale of 1 - 10 (CR10 Borg Scale) during each 60 s break within the simulated fencing bout protocol and between each simulated fencing bout.
Rating of perceived exertion of the legs | From baseline to completion, up to 31 days
  Change from baseline in rating of perceived exertion for the legs will be recorded on a scale of 1 - 10 (CR10 Borg Scale) during each 60 s break within the simulated fencing bout protocol and between each simulated fencing bout.
Rating of whole body perceived exertion | From baseline to completion, up to 31 days
  Change from baseline in whole body rating of perceived exertion will be recorded on a scale of 1 - 10 (CR10 Borg Scale) during each 60 s break within the simulated fencing bout protocol and between each simulated fencing bout.

IPD SHARING:
Plan to Share IPD: No